CLINICAL TRIAL: NCT03230292
Title: A Multicenter, 48-week, Open-label Extension Study to Assess the Long-term Safety, Tolerability, and Efficacy of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis.
Brief Title: A Study to Evaluate the Long-term Safety, Tolerability and Efficacy of Bimekizumab in Adult Patients With Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS0018; 2016-002934-57 (EudraCT Number)
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-03

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Psoriasis; Chronic Plaque Psoriasis; Bimekizumab
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Subjects in this cohort will receive dose 1 every four weeks (Q4W) subcutaneously (sc) during the 48-week open-label Treatment Period. There will be an option to increase the dose to dose 2 Q4W at the discretion of the Investigator if the subject's Psoriasis Area and Severity Index (PASI) response is >=50% to <75% reduction from the Baseline of PS0016 at Week 12 or later. If the subject's disease is adequately controlled on dose 2 Q4W, they may return to dose 1 Q4W at the discretion of the Investigator.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab will be administered subcutaneously in 2 different doses.
  Other Names: UCB4940

SUMMARY:
This is a study to assess the long-term safety, tolerability, and efficacy of bimekizumab.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have completed all dosing requirements in PS0016 without meeting any withdrawal criteria
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception up till 20 weeks after last administration of study drug, and have a negative pregnancy test at Visit 1 (Screening) and immediately prior to first dose
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active, up till 20 weeks after the last administration of study medication (anticipated 5 half-lives)

Exclusion Criteria:

* Subjects previously participating in this study
* Subject has any medical or psychiatric condition that, in the opinion of the Investigator, could jeopardize or would compromise the subject's ability to participate in this study. Note: For any subject with an ongoing serious adverse event (SAE), or a history of serious infections (including herpes zoster or hospitalizations) in PS0016, the Medical Monitor must be consulted prior to the subject's entry into PS0018
* Subject has any current sign or symptom that may indicate a medically significant infection
* Subject has current clinically active infection with Histoplasma, Coccidiodes, Paracoccidioides, Pneumocystis, tuberculosis (TB), nontuberculous mycobacteria (NTMB),Blastomyces, Aspergillus, or Candidiasis (systemic). Any subject diagnosed with Histoplasmosis, Coccidiodes, Paracoccidioides, Pneumocystis, TB, NTMB, Blastomyces, Aspergillus, or Candidiasis (systemic) during PS0016 is excluded from PS0018 even if treatment has been completed.
* Any subject who meets any withdrawal criteria in the feeder study (PS0016) is excluded from participating in the open-label extension study (PS0018)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (001 844 599 2273)
Locations (10):
- United States (2):
  - Ps0018 701, High Point, North Carolina
  - Ps0018 704, Bexley, Ohio
- Australia (4):
  - Ps0018 101, Carlton
  - Ps0018 103, East Melbourne
  - Ps0018 102, Kogarah
  - Ps0018 104, Woolloongabba
- Canada (3):
  - Ps0018 201, Ajax
  - Ps0018 203, London
  - Ps0018 202, Windsor
- Ps0018 501, Chisinau, Moldova

REFERENCES:
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- See also: Product Information — https://www.ema.europa.eu/en/documents/product-information/bimzelx-epar-product-information_en.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in July 2017 and concluded in March 2019.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- BKZ All Participants: Participants received bimekizumab (BKZ) 160 milligrams (mg) every 4 weeks (Q4W) subcutaneously (sc) during the 48-week Open Label Treatment Period. The Investigator could increase the dose to BKZ 320 mg Q4W if the participant's Psoriasis Area and Severity Index (PASI) response was greater than or equal to (>=) 50% to less than (<) 75% reduction from the Baseline of PS0016 at Week 12 or later. If the participant's disease was adequately controlled on BKZ 320 mg Q4W, they could return to BKZ 160 mg Q4W at the discretion of the Investigator.
Period: Overall Study
Arm/Group | BKZ All Participants
Started | 43
Completed | 37
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all study participants who received at least 1 dose of investigational medicinal product (IMP) in PS0018.
Arm/Group | BKZ All Participants
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 1
  White | 37

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Emergent Adverse Event (TEAE) Adjusted by Duration of Participant Exposure to Treatment
Description: TEAEs were events that had a start date on or after the first administration of study treatment in PS0018 until the last received dose of investigational medicinal product (IMP) +140 days [which covered the 20-week Safety Follow-Up (SFU) Visit]. The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that it provides an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the adverse event (AE) being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline (Week 0) until Safety Follow Up Visit (up to Week 64)
Population: The Safety Set consisted of all participants who received at least 1 dose of the study medication in PS0018.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- BKZ All Participants (SS): Participants received BKZ 160 mg Q4W sc during the 48-week Open Label Treatment Period. The Investigator could increase the dose to BKZ 320mg Q4W if the participant's PASI response was >= 50% to < 75% reduction from the Baseline of PS0016 at Week 12 or later. If the participant's disease was adequately controlled on BKZ 320 mg Q4W, they could return to BKZ 160 mg Q4W at the discretion of the Investigator. Participants formed the Safety Set (SS).
Arm/Group | BKZ All Participants (SS)
Number analyzed (Participants) | 43
no. of new events per 100 subject-years | 76.00 [53.8 to 104.3]

2. Secondary Outcome: Plasma Concentration of Bimekizumab During the Study
Description: Plasma concentration of Bimekizumab was expressed in micrograms per milliliter (μg/mL). Values Below Limit of Quantification (BLQ) were replaced by value of Lower Limit of Quantification (LLOQ) divided by 2 (=0.075 μg/mL) in calculations of Means and Coefficient of Variations (CVs). Means and CVs were only calculated if at least 2/3 of the concentrations were quantified at the respective timepoint.
Time Frame: From Baseline (Week 0) until Safety Follow Up Visit (up to Week 64)
Population: The Pharmacokinetics Per-Protocol Set consisted of all enrolled participants who received at least 1 dose of the study medication and provided at least 1 quantifiable plasma concentration postdose in PS0018. Here, 'number analyzed' signifies participants who were evaluable at specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Groups:
- BKZ All Participants (PK-PPS): Participants received BKZ 160 mg Q4W sc during the 48-week Open Label Treatment Period. The Investigator could increase the dose to BKZ 320 mg Q4W if the participant's PASI response was >= 50% to < 75% reduction from the Baseline of PS0016 at Week 12 or later. If the participant's disease was adequately controlled on BKZ 320 mg Q4W, they could return to BKZ 160 mg Q4W at the discretion of the Investigator. Participants formed the Pharmacokinetic-Per Protocol Set (PK-PPS).
Arm/Group | BKZ All Participants (PK-PPS)
Number analyzed (Participants) | 43
μg/mL
  PS0018 Week 0 | NA (NA) — Participants had no prior BKZ treatment and thus no BKZ levels at Baseline.
  Week 4: number analyzed (Participants) | 42
  Week 4 | 5.309 (47.8)
  Week 8: number analyzed (Participants) | 40
  Week 8 | 7.304 (60.7)
  Week 12: number analyzed (Participants) | 39
  Week 12 | 7.994 (53.9)
  Week 16: number analyzed (Participants) | 37
  Week 16 | 8.700 (53.7)
  Week 28: number analyzed (Participants) | 37
  Week 28 | 9.285 (49.7)
  Week 40: number analyzed (Participants) | 36
  Week 40 | 9.238 (51.3)
  Week 48/ Withdrawal: number analyzed (Participants) | 36
  Week 48/ Withdrawal | 9.056 (52.5)
  Follow-up: number analyzed (Participants) | 35
  Follow-up | 0.310 (164.8)

3. Secondary Outcome: Percentage of Participants With Positive Anti-bimekizumab (BZK) Antibody Levels Prior to Study Treatment
Description: For a given visit / time point, an Anti-BKZ status of positive was concluded for any participant with an anti-drug antibody (ADA) level that was above cut point (ACP) and CP at that visit/ time point. A participant was classified as overall positive if at least one PS0018 measurement is ACP and CP (this included participants who had negative results at PS0016 Baseline). Percentages were based on the number of participants with a non-missing measurement, from samples that did not contain BKZ concentration levels above the drug tolerance, at the visit. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: Baseline of study PS0016 [NCT03025542]
Population: The Safety Set consisted of all participants who received at least 1 dose of the study medication in PS0018.
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (SS)
Number analyzed (Participants) | 43
percentage of participants | 2.3

4. Secondary Outcome: Percentage of Participants With Overall Positive Anti-bimekizumab (BZK) Antibody Levels Following Study Treatment
Description: as for outcome 3
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: The Safety Set consisted of all participants who received at least 1 dose of the study medication in PS0018. The number of participants analyzed reflects participants with a non-missing measurement.
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (SS)
Number analyzed (Participants) | 39
percentage of participants | 25.6

5. Secondary Outcome: Percentage of Participants Achieving a 50% or Higher Improvement in Psoriasis Area and Severity Index (PASI) During the Study
Description: The PASI quantifies the severity and extent of the disease and weighs these with the percentage of body surface area (BSA) involvement. The degree of involvement is estimated across 4 body areas; head, upper limbs, trunk, and lower limbs and then transferred into a grade. The Investigator assessed the average redness, thickness, and scaliness of lesions in each body area (each on a 5 - point scale); 0 = none, 1 = slight, 2 = moderate, 3 = marked, and 4 = very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity. The PASI50 responses were based on at least 50% improvement in the PASI score at the Baseline of PS0016. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: The Full Analysis Set consisted of all enrolled participants who received at least 1 dose of the study medication and had a valid efficacy measurement for PASI at Baseline of PS0018.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- BKZ All Participants (FAS): Participants received BKZ 160 mg Q4W sc during the 48-week Open Label Treatment Period. The Investigator could increase the dose to BKZ 320 mg Q4W if the participant's PASI response was >= 50% to < 75% reduction from the Baseline of PS0016 at Week 12 or later. If the participant's disease was adequately controlled on BKZ 320 mg Q4W, they could return to BKZ 160 mg Q4W at the discretion of the Investigator. Participants formed the Full Analysis Set (FAS).
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 60.5 [45.6 to 73.6]
  Week 4 | 95.3 [84.5 to 98.7]
  Week 8 | 95.3 [84.5 to 98.7]
  Week 12 | 95.3 [84.5 to 98.7]
  Week 16 | 97.7 [87.9 to 99.6]
  Week 20 | 95.3 [84.5 to 98.7]
  Week 24 | 93.0 [81.4 to 97.6]
  Week 28 | 93.0 [81.4 to 97.6]
  Week 32 | 90.7 [78.4 to 96.3]
  Week 36 | 90.7 [78.4 to 96.3]
  Week 40 | 88.4 [75.5 to 94.9]
  Week 44 | 90.7 [78.4 to 96.3]
  Week 48/ Withdrawal | 88.4 [75.5 to 94.9]
  Follow-Up | 79.1 [64.8 to 88.6]

6. Secondary Outcome: Percentage of Participants Achieving a 75% or Higher Improvement in Psoriasis Area and Severity Index (PASI) During the Study
Description: The PASI quantifies the severity and extent of the disease and weighs these with the percentage of body surface area (BSA) involvement. The degree of involvement is estimated across 4 body areas; head, upper limbs, trunk, and lower limbs and then transferred into a grade. The Investigator assessed the average redness, thickness, and scaliness of lesions in each body area (each on a 5 - point scale); 0 = none, 1 = slight, 2 = moderate, 3 = marked, and 4 = very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity. The PASI75 responses were based on at least 75% improvement in the PASI score at the Baseline of PS0016. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 44.2 [30.4 to 58.9]
  Week 4 | 88.4 [75.5 to 94.9]
  Week 8 | 95.3 [84.5 to 98.7]
  Week 12 | 90.7 [78.4 to 96.3]
  Week 16 | 93.0 [81.4 to 97.6]
  Week 20 | 90.7 [78.4 to 96.3]
  Week 24 | 90.7 [78.4 to 96.3]
  Week 28 | 88.4 [75.5 to 94.9]
  Week 32 | 90.7 [78.4 to 96.3]
  Week 36 | 90.7 [78.4 to 96.3]
  Week 40 | 86.0 [72.7 to 93.4]
  Week 44 | 90.7 [78.4 to 96.3]
  Week 48/ Withdrawal | 86.0 [72.7 to 93.4]
  Follow-Up | 65.1 [50.2 to 77.6]

7. Secondary Outcome: Percentage of Participants Achieving a 90% or Higher Improvement in Psoriasis Area and Severity Index (PASI) During the Study
Description: The PASI quantifies the severity and extent of the disease and weighs these with the percentage of body surface area (BSA) involvement. The degree of involvement is estimated across 4 body areas; head, upper limbs, trunk, and lower limbs and then transferred into a grade. The Investigator assessed the average redness, thickness, and scaliness of lesions in each body area (each on a 5 - point scale); 0 = none, 1 = slight, 2 = moderate, 3 = marked, and 4 = very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity. The PASI90 responses were based on at least 90% improvement in the PASI score at the Baseline of PS0016. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 20.9 [11.4 to 35.2]
  Week 4 | 53.5 [38.9 to 67.5]
  Week 8 | 79.1 [64.8 to 88.6]
  Week 12 | 79.1 [64.8 to 88.6]
  Week 16 | 86.0 [72.7 to 93.4]
  Week 20 | 79.1 [64.8 to 88.6]
  Week 24 | 79.1 [64.8 to 88.6]
  Week 28 | 81.4 [67.4 to 90.3]
  Week 32 | 81.4 [67.4 to 90.3]
  Week 36 | 86.0 [72.7 to 93.4]
  Week 40 | 76.7 [62.3 to 86.8]
  Week 44 | 86.0 [72.7 to 93.4]
  Week 48/ Withdrawal | 79.1 [64.8 to 88.6]
  Follow-Up | 58.1 [43.3 to 71.6]

8. Secondary Outcome: Percentage of Participants Achieving a 100% Improvement in Psoriasis Area and Severity Index (PASI) During the Study
Description: The PASI quantifies the severity and extent of the disease and weighs these with the percentage of body surface area (BSA) involvement. The degree of involvement is estimated across 4 body areas; head, upper limbs, trunk, and lower limbs and then transferred into a grade. The Investigator assessed the average redness, thickness, and scaliness of lesions in each body area (each on a 5 - point scale); 0 = none, 1 = slight, 2 = moderate, 3 = marked, and 4 = very marked. The PASI score ranges from 0 to 72 with a higher score indicating increased disease severity. The PASI100 responses were based on 100% improvement in the PASI score at the Baseline of PS0016. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 4.7 [1.3 to 15.5]
  Week 4 | 23.3 [13.2 to 37.7]
  Week 8 | 37.2 [24.4 to 52.1]
  Week 12 | 46.5 [32.5 to 61.1]
  Week 16 | 39.5 [26.4 to 54.4]
  Week 20 | 48.8 [34.6 to 63.2]
  Week 24 | 41.9 [28.4 to 56.7]
  Week 28 | 46.5 [32.5 to 61.1]
  Week 32 | 41.9 [28.4 to 56.7]
  Week 36 | 41.9 [28.4 to 56.7]
  Week 40 | 46.5 [32.5 to 61.1]
  Week 44 | 46.5 [32.5 to 61.1]
  Week 48/ Withdrawal | 46.5 [32.5 to 61.1]
  Follow-Up | 18.6 [9.7 to 32.6]

9. Secondary Outcome: Percentage of Participants With Investigator´s Global Assessment (IGA) Response (Clear or Almost Clear With at Least a 2 Category Improvement From Baseline on a 5-point Scale) During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0=Clear to 4=Severe. The response was defined as clear [0] or almost clear [1] with at least 2 category improvement from PS0016 Baseline. Clear was defined as no signs of PSO; post-inflammatory hyperpigmentation may be present. Almost clear was defined as no thickening; normal to pink coloration; no to minimal focal scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: The Full Analysis Set consisted of all enrolled participants who received at least 1 dose of the study medication and have a valid efficacy measurement for PASI at Baseline of PS0018.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 18.6 [9.7 to 32.6]
  Week 4 | 62.8 [47.9 to 75.6]
  Week 8 | 79.1 [64.8 to 88.6]
  Week 12 | 79.1 [64.8 to 88.6]
  Week 16 | 81.4 [67.4 to 90.3]
  Week 20 | 79.1 [64.8 to 88.6]
  Week 24 | 76.7 [62.3 to 86.8]
  Week 28 | 79.1 [64.8 to 88.6]
  Week 32 | 86.0 [72.7 to 93.4]
  Week 36 | 81.4 [67.4 to 90.3]
  Week 40 | 79.1 [64.8 to 88.6]
  Week 44 | 83.7 [70.0 to 91.9]
  Week 48/ Withdrawal | 79.1 [64.8 to 88.6]
  Follow-Up | 51.2 [36.8 to 65.4]

10. Secondary Outcome: Mean Change From PS0016 [NCT03025542] Baseline in PASI Score During the Study
Description: The total PASI score ranges from 0 to 72 with a reduction from PS0016 Baseline indicating improvement. Missing data was imputed using Last observation carried forward (LOCF) at all visits. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
score on a scale
  PS0018 Week 0 | -11.21 (9.13)
  Week 4 | -16.79 (6.72)
  Week 8 | -18.12 (7.41)
  Week 12 | -18.70 (7.89)
  Week 16 | -19.01 (8.70)
  Week 20 | -18.91 (8.70)
  Week 24 | -19.08 (8.66)
  Week 28 | -19.13 (8.79)
  Week 32 | -19.30 (8.66)
  Week 36 | -19.27 (8.68)
  Week 40 | -19.22 (8.82)
  Week 44 | -19.32 (8.68)
  Week 48/ Withdrawal | -19.20 (8.76)
  Follow-up | -15.93 (9.29)

11. Secondary Outcome: Mean Percentage Change From PS0016 [NCT03025542] Baseline in PASI Score During the Study
Description: A negative percentage change from PS0016 baseline indicated improvement in Total PASI score. The total PASI score ranges from 0 to 72 with a reduction from PS0016 Baseline indicating improvement. Missing data was imputed using Last Observation Carried Forward (LOCF) at all visits. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage change
  PS0018 Week 0 | -56.45 (38.26)
  Week 4 | -87.71 (15.52)
  Week 8 | -93.28 (12.13)
  Week 12 | -94.50 (8.22)
  Week 16 | -95.15 (8.43)
  Week 20 | -94.84 (9.02)
  Week 24 | -95.69 (6.77)
  Week 28 | -95.72 (7.35)
  Week 32 | -96.85 (4.81)
  Week 36 | -96.66 (4.88)
  Week 40 | -96.13 (6.38)
  Week 44 | -96.98 (4.14)
  Week 48/ Withdrawal | -96.10 (7.45)
  Follow-Up | -81.98 (25.45)

12. Secondary Outcome: Percentage of Participants Who Shifted From Moderate Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Clear IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Moderate IGA was defined as clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling. Clear IGA was defined as no signs of PSO; post-inflammatory hyperpigmentation may be present. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 4.7
  Week 4 | 23.3
  Week 8 | 37.2
  Week 12 | 44.2
  Week 16 | 34.9
  Week 20 | 41.9
  Week 24 | 37.2
  Week 28 | 39.5
  Week 32 | 37.2
  Week 36 | 37.2
  Week 40 | 37.2
  Week 44 | 37.2
  Week 48/ Withdrawal | 39.5
  Follow-Up | 18.6

13. Secondary Outcome: Percentage of Participants Who Shifted From Moderate Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Almost Clear IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Moderate IGA was defined as clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling. Almost clear was defined as no thickening; normal to pink coloration; no to minimal focal scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 11.6
  Week 4 | 37.2
  Week 8 | 32.6
  Week 12 | 23.3
  Week 16 | 37.2
  Week 20 | 23.3
  Week 24 | 30.2
  Week 28 | 30.2
  Week 32 | 37.2
  Week 36 | 30.2
  Week 40 | 27.9
  Week 44 | 32.6
  Week 48/ Withdrawal | 25.6
  Follow-Up | 30.2

14. Secondary Outcome: Percentage of Participants Who Shifted From Moderate Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Mild IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Moderate IGA was defined as clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling. Mild was defined as just detectable to mild thickening; pink to light red coloration; predominately fine scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 25.6
  Week 4 | 18.6
  Week 8 | 14.0
  Week 12 | 11.6
  Week 16 | 9.3
  Week 20 | 14.0
  Week 24 | 9.3
  Week 28 | 7.0
  Week 32 | 2.3
  Week 36 | 9.3
  Week 40 | 9.3
  Week 44 | 2.3
  Week 48/ Withdrawal | 7.0
  Follow-Up | 11.6

15. Secondary Outcome: Percentage of Participants Who Shifted From Moderate Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Moderate IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Moderate IGA was defined as clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 25.6
  Week 4 | 4.7
  Week 8 | 0
  Week 12 | 2.3
  Week 16 | 2.3
  Week 20 | 2.3
  Week 24 | 2.3
  Week 28 | 2.3
  Week 32 | 0
  Week 36 | 0
  Week 40 | 2.3
  Week 44 | 4.7
  Week 48/ Withdrawal | 4.7
  Follow-Up | 11.6

16. Secondary Outcome: Percentage of Participants Who Shifted From Moderate Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Severe IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Moderate IGA was defined as clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling. Severe was defined as severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 16.3
  Week 4 | 0
  Week 8 | 0
  Week 12 | 0
  Week 16 | 0
  Week 20 | 0
  Week 24 | 0
  Week 28 | 0
  Week 32 | 0
  Week 36 | 0
  Week 40 | 0
  Week 44 | 0
  Week 48/ Withdrawal | 0
  Follow-Up | 4.7

17. Secondary Outcome: Percentage of Participants Who Shifted From Severe Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Clear IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Severe IGA was defined as severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. Clear was defined as no signs of PSO; post-inflammatory hyperpigmentation may be present. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 0
  Week 4 | 0
  Week 8 | 0
  Week 12 | 2.3
  Week 16 | 4.7
  Week 20 | 7.0
  Week 24 | 4.7
  Week 28 | 7.0
  Week 32 | 4.7
  Week 36 | 7.0
  Week 40 | 11.6
  Week 44 | 9.3
  Week 48/ Withdrawal | 9.3
  Follow-Up | 0

18. Secondary Outcome: Percentage of Participants Who Shifted From Severe Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Almost Clear IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Severe IGA was defined as severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. Almost clear was defined as no thickening; normal to pink coloration; no to minimal focal scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 2.3
  Week 4 | 2.3
  Week 8 | 9.3
  Week 12 | 9.3
  Week 16 | 4.7
  Week 20 | 7.0
  Week 24 | 4.7
  Week 28 | 2.3
  Week 32 | 7.0
  Week 36 | 7.0
  Week 40 | 2.3
  Week 44 | 4.7
  Week 48/ Withdrawal | 4.7
  Follow-Up | 2.3

19. Secondary Outcome: Percentage of Participants Who Shifted From Severe Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Mild IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Severe IGA was defined as severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. Mild was defined as just detectable to mild thickening; pink to light red coloration; predominately fine scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 2.3
  Week 4 | 9.3
  Week 8 | 2.3
  Week 12 | 0
  Week 16 | 4.7
  Week 20 | 0
  Week 24 | 4.7
  Week 28 | 4.7
  Week 32 | 2.3
  Week 36 | 0
  Week 40 | 0
  Week 44 | 0
  Week 48/ Withdrawal | 0
  Follow-Up | 7.0

20. Secondary Outcome: Percentage of Participants Who Shifted From Severe Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Moderate IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Severe IGA was defined as severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. Moderate was defined as clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 2.3
  Week 4 | 2.3
  Week 8 | 0
  Week 12 | 2.3
  Week 16 | 0
  Week 20 | 0
  Week 24 | 0
  Week 28 | 0
  Week 32 | 0
  Week 36 | 0
  Week 40 | 0
  Week 44 | 0
  Week 48/ Withdrawal | 0
  Follow-Up | 2.3

21. Secondary Outcome: Percentage of Participants Who Shifted From Severe Investigator´s Global Assessment (IGA) Score at PS0016 [NCT03025542] Baseline to Severe IGA Score During the Study
Description: A static IGA for Psoriasis (PSO) was used to assess disease severity in all study participants during the study. IGA is a 5 point scale ranging from 0 = Clear to 4 = Severe. Severe IGA was defined as severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0018 Week 0 | 9.3
  Week 4 | 2.3
  Week 8 | 2.3
  Week 12 | 0
  Week 16 | 0
  Week 20 | 0
  Week 24 | 0
  Week 28 | 0
  Week 32 | 0
  Week 36 | 0
  Week 40 | 0
  Week 44 | 0
  Week 48/ Withdrawal | 0
  Follow-Up | 2.3

22. Secondary Outcome: Mean Percentage in the Body Surface Area (BSA) Affected by Psoriasis During the Study
Description: The BSA palm method was used for the evaluation of BSA as follows: Body surface area estimation used the palm (study participant's flat hand and thumb together, fingers included) as representing around 1% of the total BSA. Missing data was imputed using Last Observation Carried forward (LOCF) at all visits. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of BSA
  PS0016 Baseline | 25.8 (17.5)
  PS0018 Week 0 | 8.6 (10.7)
  Week 4 | 5.2 (12.6)
  Week 8 | 3.0 (10.9)
  Week 12 | 2.0 (4.8)
  Week 16 | 1.0 (1.6)
  Week 20 | 1.2 (2.2)
  Week 24 | 1.2 (1.9)
  Week 28 | 0.9 (1.6)
  Week 32 | 0.8 (1.1)
  Week 36 | 0.7 (1.1)
  Week 40 | 0.8 (1.2)
  Week 44 | 0.7 (1.0)
  Week 48/ Withdrawal | 0.7 (1.2)
  Follow-Up | 4.8 (13.0)

23. Secondary Outcome: Mean Percentage Change From PS0016 [NCT03025542] Baseline in the Body Surface Area (BSA) Affected by Psoriasis During the Study
Description: The percentage BSA (0 to 100%) affected by PSO was listed by PS0016 randomized treatment, by study participant and visit including the percentage change from PS0016 Baseline. The BSA palm method was used for the evaluation of BSA as follows: Body surface area estimation used the palm (study participant's flat hand and thumb together, fingers included) as representing around 1% of the total BSA. Missing data was imputed using Last observation carried forward (LOCF) at all visits. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: From Baseline of study PS0016 [NCT03025542] until Safety Follow Up Visit (up to Week 64) of study PS0018
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage change
  PS0018 Week 0 | -61.0 (41.5)
  Week 4 | -83.0 (23.7)
  Week 8 | -91.1 (15.9)
  Week 12 | -92.9 (10.9)
  Week 16 | -95.5 (7.4)
  Week 20 | -94.4 (9.1)
  Week 24 | -94.8 (7.8)
  Week 28 | -95.4 (8.7)
  Week 32 | -96.1 (6.7)
  Week 36 | -96.5 (5.7)
  Week 40 | -95.8 (8.5)
  Week 44 | -96.3 (6.2)
  Week 48/ Withdrawal | -95.6 (10.0)
  Follow-Up | -81.5 (33.9)

24. Secondary Outcome: Mean Change From PS0016 [NCT03025542] Baseline in Hospital Anxiety and Depression Scale - Anxiety (HADS-A) Score During the Study
Description: HADS-A score is the sum of the 7 individual scores in the anxiety domain and ranges from 0 to 21 with higher scores indicating worse state. A score below 8 was considered normal whereas a score of 15 and above was considered severe. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: Week 0, 12, 24, 36, and 48 of study PS0018, Relative to Baseline of study PS0016 [NCT03025542]
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
score on a scale
  PS0018 Week 0 | -1.5 (2.3)
  Week 12 | -2.0 (1.8)
  Week 24 | -2.0 (2.4)
  Week 36 | -2.0 (2.4)
  Week 48/ Withdrawal | -1.5 (2.2)

25. Secondary Outcome: Mean Change From PS0016 [NCT03025542] Baseline in Hospital Anxiety and Depression Scale - Depression (HADS-D) Score During the Study
Description: HADS-D score is the sum of the 7 individual scores in the depression domain and ranges from 0 to 21 with higher scores indicating worse state. A score below 8 was considered normal whereas a score of 15 and above was considered severe. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: Week 0, 12, 24, 36, and 48 of study PS0018, Relative to Baseline of study PS0016 [NCT03025542]
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
score on a scale
  PS0018 Week 0 | -1.0 (1.4)
  Week 12 | -0.8 (2.1)
  Week 24 | -1.0 (1.7)
  Week 36 | -1.1 (1.7)
  Week 48/ Withdrawal | -1.0 (1.8)

26. Secondary Outcome: Percentage of Participants With Scores Below 8 in HADS-A (Participants With Normal Scores) During the Study
Description: HADS-A score is the sum of the 7 individual scores in the anxiety domain and ranges from 0 to 21 with higher scores indicating worse state. A score below 8 was considered normal. Percentages were based on the number of participants with a non-missing measurement at the visit. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: Baseline of study PS0016 [NCT03025542], Week 0, 12, 24, 36, and 48 of study PS0018
Population: The Full Analysis Set consisted of all enrolled participants who received at least 1 dose of the study medication and have a valid efficacy measurement for PASI at Baseline of PS0018. Here, 'number analyzed' signifies participants who were evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0016 Baseline | 83.7
  PS0018 Week 0 | 88.4
  Week 12: number analyzed (Participants) | 42
  Week 12 | 95.2
  Week 24: number analyzed (Participants) | 42
  Week 24 | 90.5
  Week 36: number analyzed (Participants) | 39
  Week 36 | 89.7
  Week 48/ Withdrawal: number analyzed (Participants) | 39
  Week 48/ Withdrawal | 87.2

27. Secondary Outcome: Percentage of Participants With Scores Below 8 in HADS-D (Participants With Normal Scores) During the Study
Description: HADS-D score is the sum of the 7 individual scores in the depression domain and ranges from 0 to 21 with higher scores indicating worse state. A score below 8 was considered normal. Percentages were based on the number of participants with a non-missing measurement at the visit. Baseline was defined as the last available value prior to the first injection of study medication in the PS0016 study.
Time Frame: Baseline of study PS0016 [NCT03025542], Week 0, 12, 24, 36, and 48 of study PS0018
Population: as for outcome 26
Measure: Number; unit: percentage of participants
Arm/Group | BKZ All Participants (FAS)
Number analyzed (Participants) | 43
percentage of participants
  PS0016 Baseline | 93.0
  PS0018 Week 0 | 97.7
  Week 12: number analyzed (Participants) | 42
  Week 12 | 95.2
  Week 24: number analyzed (Participants) | 42
  Week 24 | 97.6
  Week 36: number analyzed (Participants) | 39
  Week 36 | 94.9
  Week 48/ Withdrawal: number analyzed (Participants) | 39
  Week 48/ Withdrawal | 97.4

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the PS0018 Baseline until the Safety Follow-Up Visit [20 weeks after the last dose (up to Week 64)]
Arm/Group | BKZ All Participants (SS)
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 3/43
Other Adverse Events (participants affected / at risk) | 27/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BKZ All Participants (SS) (N=43)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BKZ All Participants (SS) (N=43)
Upper respiratory tract infection (Infections and infestations) | 8 (12)
Nasopharyngitis (Infections and infestations) | 7 (10)
Viral upper respiratory tract infection (Infections and infestations) | 5 (6)
Oral candidiasis (Infections and infestations) | 4 (6)
Pharyngitis (Infections and infestations) | 3 (3)
Staphylococcal pharyngitis (Infections and infestations) | 3 (3)
Gamma-glutamyltransferase increased (Investigations) | 5 (7)
Alanine aminotransferase increased (Investigations) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03230292/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT03230292/SAP_001.pdf